CLINICAL TRIAL: NCT03221322
Title: The Investigation of Lifestyle and Genetics in Super Lean Subjects That Keep Them Resistant to Weight Gain
Brief Title: How do Super Lean Subjects Keep Resistant to Body Weight Gain?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sumei Hu, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: 0060
Record Dates: First submitted 2017-06-27; First posted 2017-07-18 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Thinness; Health Behavior; Genetics
MeSH Terms: conditions — Thinness; Health Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 9 ml of blood samples will be collected for the biological measurements and DNA extraction for genotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: 20 kg/m2 ≤ BMI ≤ 25 kg/m2, healthy, with no eating disorder, 150 subjects, 20 - 40 years old
  Interventions: Behavioral: Superlean
- Superlean: 15 kg/m2 ≤ BMI ≤ 18 kg/m2, healthy, with no eating disorder, 150 subjects, 25 - 35 years old in particular
  Interventions: Behavioral: Superlean

INTERVENTIONS:
Behavioral: Superlean — Behavioural data will be collected on all subjects in either control group or superlean group. Blood or saliva samples will be collected for DNA extraction and genotyping.

SUMMARY:
Obesity is the 5th leading cause of global death, and is major risk factors for many chronic diseases, such as type 2 diabetes, cardiovascular diseases, hypertension and cancer. Obesity is caused by an imbalance between energy intake and energy expenditure, and it is widely agreed to be a consequence of a gene by environment interaction. Although on average obesity rates are increasing, the shape of the distribution of adiposity is changing: it is becoming more right skewed. This is because there is a population of very lean subjects that has remained almost unchanged by the epidemic. The investigators have called these very lean individuals that are resistant to the epidemic and sustain a BMI < 18.5 kg/m2 'super lean' subjects. We have very little understanding of the lifestyles of these individuals and how they are able to maintain their super lean phenotype, and whether the basis of their leanness is primarily genetics.

DETAILED DESCRIPTION:
In this study, the investigators will recruit a sample of 150 super lean healthy volunteers with a BMI >15 and < 18.5 kg/m2 aged 20-40 years, in parallel with an age matched group of 150 healthy subjects with a BMI ≥22 and < 25 kg/m2 as the control group. The investigators will screen out any individuals with eating disorders. In both groups, the investigators will study their lifestyles in particular focusing on their physical activity patterns and their food intake choices (monitored via food intake diaries and supported by metabolomics analyses of their urine to detect biomarkers of different food groups). Saliva samples will be collected for genotyping. The investigators will SNP genotype the individuals for 30 known polymorphic loci previously linked to obesity to establish if they have a particular genetic profile linked to their lean phenotype.

ELIGIBILITY:
Inclusion Criteria:

* control: BMI 20-25 kg/m2, healthy, age 20-40 years old superlean: BMI 15-18 kg/m2, healthy, with no eating disorders and diabetes, age 20-40 years old

Exclusion Criteria:

* Pregnant women and women in lactation Subjects are suffering from eating disorders or diabetes.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are healthy, with no eating disorder, 25 - 35 years old in particular.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurements of participants in both control and superlean groups | Through study completion, an average of 2 years
  Height, waist and hip circumferences (cm) and body composition will be measured on arrival.
Demographic characteristics of all participants in both control and superlean groups | Through study completion, an average of 2 years
  Life style questionnaire filled out on arrival.

CONTACTS AND LOCATIONS:
Overall Officials: John Speakman, PhD, Principal Investigator — Institute of Genetics and Developmental Biology
Locations (1):
- Institute of Genetics and Developmental Biology, Beijing, China

IPD SHARING:
Plan to Share IPD: No